CLINICAL TRIAL: NCT05953025
Title: The Effect of Short Term Continuous Positive Airway Pressure Treatment on Depressive Symptoms in Obstructive Sleep Apnoea Syndrome Patients, Including Anti-depressant Treatment Resistant Patients: An Observational Study
Brief Title: Obersvational Study on Effects of CPAP on Depressive Symptoms in OSAS
Acronym: COAST
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2017/65
Record Dates: First submitted 2023-04-06; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — No intervention on care- questionnaire to see effect of standard care treatment on symptoms

SUMMARY:
The official definition of depression or major depressive disorder, is a psychological disorder which is characterised by a persistent low mood or loss of interest in previously pleasurable activities, for over two weeks. It is one of the leading causes of disability world-wide and is one of the most common mental health disorders, affecting 5-10% of the world population at any one time. However, a major problem with this condition is the over-use of antidepressants. The number of anti-depressant prescriptions has doubled in the last decade and cost the NHS £780,000 per day in 2015.

Many of the symptoms of obstructive sleep apnoea syndrome (OSAS) are similar to symptoms of depression, such as fatigue, low mood, difficulty concentrating and un-refreshing sleep. This means that patients could be misdiagnosed with depression and begin on courses of antidepressants which don't improve their symptoms.

A very high association between OSAS and depression has been consistently recorded in research studies. Similarly, the primary treatment for OSAS, continuous positive airway pressure (CPAP) has been shown to significantly improve depressive symptoms in these patients. However, when studying the effects CPAP therapy has on patients with OSAS, one of the main factors which can cause differences is in antidepressant use. A lot of studies have excluded those who are on them, while quite a lot failed to note the antidepressant use. Therefore, this study aims to focus on those patients who are on antidepressant therapy but not gaining remission in their symptoms. These patients may be classed as anti-depressant treatment resistant.

DETAILED DESCRIPTION:
4.2 Participant Role

The study will be an observational study, using questionnaires at three time points. The first will be when the participant attends their initial sleep consultation. If the participant's symptoms are indicative of OSAS, they will be sent for a home sleep study. If this is diagnostic for OSAS, the participant will begin their treatment with CPAP and attend a follow up 6-8 weeks after that, to review their treatment. The second and third times will be at these two appointments. The questionnaires used will be:

* Baseline demographic data - used to gain information about the participant.
* The Patient Health Questionnaire 9 - used to quantify the patient's depressive symptoms.
* The Massachusetts General Hospital - Antidepressant treatment resistant questionnaire - used to quantify if a patient is antidepressant treatment resistant.
* The Epworth Sleepiness Scale - used to quantify how likely the patient is to fall asleep.
* The Fatigue Severity Scale - used to quantify how fatigued the patient is. The patient's OSAS severity and compliance with CPAP will also be assessed. 4.3 Study Impact As mentioned previously, the cost of antidepressants to the NHS is increasing. More studies are required to assess if there is a potential for alternative testing, before a patient begins on antidepressants. This study aims to show that patients may have been misdiagnosed with depression and that an underlying sleep problem is the cause of their symptoms. Therefore, a referral for a sleep study may be more appropriate than a prescription for antidepressants.

  5. BACKGROUND AND RATIONALE 5.1 Depression and Treatment Resistance Major depressive disorder, or depression, is a psychological disorder characterised by a persistent low mood or loss of interest in previously pleasurable activities, for over two weeks . It is one of the most prevalent mental health disorders. The World Health Organisation estimated that 5-10% of the world population are suffering with identifiable depression at any one time, while the lifetime risk of developing depression is between 10-20%. Depression also has a greater impact on health status than chronic systemic diseases, such as angina and diabetes, making it one of the leading causes of disease burden worldwide However, one of the greatest issues facing people with depression is that approximately 60% of those treated are not achieving an adequate response . These patients are classified as having treatment resistant depression (TRD). Although there is no universally accepted definition , a commonly accepted definition is a failure to respond to two or more antidepressants, given sequentially at an adequate dose for an adequate time. The prevalence of approximately 60% has been repeatedly reported in many large clinical trials, with the Sequenced Treatment Alternatives to Relive Depression trial recorded that only a third of patients responded to their initial antidepressant therapy Another study reported an 11% remission rate and 26.3% response rate following 12 months of depression treatment. This has become a growing problem for the NHS and the UK economy. The number of anti-depressant prescriptions has been continually rising, it has doubled in the last decade and cost the NHS £780,000 per day in 2015 . There is also a great cost to the patient, as the absence of remission is associated with impairment in work, social and family life, as well as increasing mortality .

5.2 Association Between Depression and Obstructive Sleep Apnoea Syndrome Obstructive sleep apnoea syndrome (OSAS) can affect people of any age, however it is most prevalent in those aged 30 to 65, being present in 4% of men and 2% of women in this age group. OSAS is characterised by excessive daytime sleepiness, with periods of >10 second partial (hypopnoea) or complete (apnoea) obstruction of the upper airway. Hypopneas/apnoeas lead to desaturation in blood oxygen levels and are accompanied by an arousal to wakefulness or light sleep, which fragments the normal sleep cycle. NICE recommend using the Epworth Sleepiness Scale (ESS) to objectively assess the patient's perception of sleepiness and the extent and severity of symptoms. OSAS is associated with impaired quality of life, cognitive dysfunction, and psychological disorders, such as anxiety and depression. Although there is heterogeneity, a significantly higher prevalence of depression among OSAS patients has been reported than in the general population. An epidemiological study of 18,980 patients in various countries across Europe found 17.6% of subjects with a previous diagnosis of OSAS, also had a diagnosis of depression. This was also supported by a retrospective study on the medical notes of approximately 4 million veterans, which reported that of the 118,105 patients with OSAS, 21.8% had comorbid depression. This was approximately 3 times higher than those without OSAS . There has been a greater prevalence reported of patients with depression and OSAS within sleep clinics, even as high as 63%. Conversely, one study reported that 63% of patients diagnosed with depression reported having sleep problems. The reason for this clinically significant association is not fully understood. It is theorised that the severe sleepiness that patients with OSAS feel, may be misinterpreted as symptoms of depression and lead to a clinical misdiagnosis. In fact, NICE recommend suspecting OSAS when patients present with symptoms of "mood swings, personality changes, or depression". Therefore, this shows that the two disorders can present similarly, and patients could be being misdiagnosed.

5.3 Continuous Positive Airway Pressure Continuous positive airway pressure (CPAP) treatment is the recommended treatment option for patients with moderate-severe OSAS. It is also recommended for those with mild OSAS if their symptoms affect their quality of life and lifestyle advice has not improved symptoms. CPAP has been shown to effectively treat OSAS, reduce excessive sleepiness and adverse events related to other medical conditions. NICE reviewed 23 randomised control trials and found CPAP caused a significant improvement in the patients' daytime sleepiness, -2.7 on the ESS, compared to placebo. CPAP is a device that generates airflow, through a facemask, nasal mask or helmet device into to the airway. This positive pressure produced by the airflow stents the airway open and prevents it collapsing in an apnoea or hypopnea . For CPAP treatment to be effective the person must wear their device when they go to sleep. Therefore, compliance is very important to the effectiveness of the device. The Portsmouth NHS Trust sleep team define compliance as the percentage of nights the patient wore their CPAP device for more than 4 hours. Ideally this should be greater than 70%.

5.4 The Effect of CPAP Depressive Symptoms A number of studies have compared the effects of CPAP treatment of OSA on depressive symptoms. A meta-analysis by Povitz et al compared 19 randomised control trials and found that CPAP treatment resulted in a significant improvement in depressive symptoms compared to control groups (p=0.004), but with significant heterogeneity between trials (p=0.001). The Patient Health Questionnaire 9 (PHQ-9) is a validated self-rating depression questionnaire that categorises depression as a score ≥10 . Edwards et al used the PHQ-9 on 293 participants undergoing 3 months of CPAP, finding a significant improvement in the patients' depressive scores, with an average decrease from 11.3±6.1 to 3.7±2.9. One of the largest methodological differences is in documentation of antidepressant use. Povitz et al, (2014) noted only 6 trials excluded participants using antidepressants and one excluded the use of benzodiazepines, but none of the others reported the use or initiation of antidepressants in their studies. As mentioned previously, antidepressant use varies a lot between different patients and therefore is an important cofounding factor. To date, only Habukawa et al (have studied the effect of CPAP treatment on depressive symptoms specifically within the TRD population. This preliminary study was in a limited sample size of 17 patients but found a significant decrease in both the self-rating Beck Depression Index and the clinician-administered Hamilton Rating Scale for Depression (both p<0.01) after 2 months of CPAP treatment. There are three major TRD classification systems, a 5-stages classification, a National Institute of Clinical Excellence (NICE) algorithm, and the Massachusetts General Hospital (MGH) criteria. The MGH produced a validated self-rated questionnaire to determine TRD, the MGH-Antidepressant Treatment Response Questionnaire (MGH-ATRQ) (Chandler et al., 2010). This will be used in the present study to assess TRD.

5.5 Conclusion Previous research has clearly shown a strong association between CPAP treatment and improvement in depressive symptoms. However, not recording patients' antidepressant use or excluding patients on antidepressants is not representative of the general population, and does not tackle the issue of TRD patients. Therefore, there is a need for more studies investigating the effects of CPAP treatment on TRD patients. The current observational study aims to build on the research performed by Habukawa et al. This will not only be done by involving a larger sample size, but also by using the MGH-ATRQ as an objective quantification of TRD. We also aim to provide more information about the behaviours of those with TRD, for example if their compliance with CPAP or self-rated sleepiness varies from other patients with OSAS. Another confounding factor could be fatigue; therefore our study will also use the validated, self-reported fatigue questionnaire, Fatigue Severity Scale (FSS) as a way to quantify any differences in patients' perception of fatigue.

The study aims to encourage further research into the area, as well as provide more evidence to persuade clinicians to refer patients for sleep studies, rather than prescribing increasing doses of antidepressants. This could have a significant benefit to clinical practice, patients' quality of lives and cost to the NHS but reducing the over-reliance on anti-depressant medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 years or above
* Be treated by the Portsmouth NHS Trust Sleep Department
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* • Has a disorder, including cognitive dysfunction, which would impair their ability to accurately complete the questionnaires or provide informed consent

  * Unable to read or understand basic English (an interpreter will not be available for this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have an appointment to attend a consultation in the sleep department of Queen Alexandra Hospital. The majority will be diagnosed with OSAS following a sleep consultation and a home sleep study. They will then be beginning a course of CPAP therapy for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptom | Over the course of the entire study- 10 months
  To assess changes in depressive symptoms of patients with OSAS at 6 weeks following CPAP treatment, using the PHQ-9 questionnaire

SECONDARY OUTCOMES:
Describe depressive symptoms | Over the course of the entire study- 10 months
  To describe depressive symptoms and changes in these for the whole cohort and in subgroups of patients, for example those with significant depressive scores (PHQ-9 ≥ 10) but not on anti-depressant medication, and "treatment resistant patients" with significant depressive scores (dependent on MGH-ATRQ) at 6 weeks, those not diagnosed with OSAS
Somnolence in the whole cohort | Over the course of the entire study- 10 months
  To describe somnolence in the whole cohort (using the ESS), and in subgroups of patients (significant depressive scores with and without treatment resistance and non-significant depressive scores, those not diagnosed with OSAS)
Describe fatigue in the cohort | Over the course of the entire study- 10 months
  To describe fatigue in the whole cohort (using FSS), and in subgroups of patients (significant depressive scores with and without treatment resistance and non-significant depressive scores, those not diagnosed with OSAS)
Describe OSAS severity | Over the course of the entire study- 10 months
  To describe OSAS severity in the whole cohort (using AHI) and in subgroups of patients (significant depressive scores with and without treatment resistance and non-significant depressive scores, those not diagnosed with OSAS)
Relationships between scores | Over the course of the entire study- 10 months [response to comment- this study has already completed using these outcome measures- no more updates to this will be made]
  Can any relationships between PHQ-9 score, FSS, ESS, likelihood and severity of OSAS, and CPAP compliance be identified?
Diagnostic differences | Over the course of the entire study- 10 months [response to comment- this study has already completed using these outcome measures- no more updates to this will be made]
  Can differences between those who are and are not diagnosed with OSAS be identified on initial presentation?

CONTACTS AND LOCATIONS:
Overall Officials: Tess Compton-Price, Principal Investigator — Lead Therapist
Locations (1):
- Portsmouth Hospitals NHS Trust, Cosham, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No